CLINICAL TRIAL: NCT04202068
Title: A Study Evaluating Efficacy and Safety of Ceftriaxone Sodium and Sulbactam Sodium for Injection in the Treatment of Uncomplicated Urogenital Gonorrhea
Brief Title: A Study Evaluating Efficacy and Safety of CRO-SBT in the Treatment of Gonorrhea
Acronym: CRO-SBT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiangbei Welman Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC0048-015
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Gonorrhea
MeSH Terms: conditions — Gonorrhea | interventions — Ceftriaxone; Sulbactam; Injections

STUDY DESIGN:
Intervention Model Description: Ceftriaxone sodium and Sulbactam Sodium for injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ceftriaxone sodium and Sulbactam Sodium for injection (Experimental): combinations of β-Lactamase inhibitors
  Interventions: Drug: Ceftriaxone sodium and Sulbactam Sodium for injection

INTERVENTIONS:
Drug: Ceftriaxone sodium and Sulbactam Sodium for injection — Ceftriaxone sodium and Sulbactam Sodium for injection is available as sterile powder for reconstitution.It will be administered as one 3g IV dose for adult or one 75mg/kg IV dose for children under 12.
  Other Names: CRO-SBT

SUMMARY:
This is a phaseIV, multicenter, open-label，single arm study which will be performed to evaluate efficacy and safety of Ceftriaxone sodium and Sulbactam Sodium for injection for the treatment of uncomplicated urogenital infection caused by Neisseria gonorrhoeae in adolescent and adult subjects.

DETAILED DESCRIPTION:
In this study, adults will be administered as one 3g IV dose at the study site,Children under 12 will be administered as one 75mg/kg IV dose . Approximately 100 subjects will be recruited to receive study treatment. The duration of the study will be approximately 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be >=6 or ≦80 years of age at the time of signing the informed consent,both gender
* Subjects having clinical suspicion of a urogenital gonococcal infection with or without gonococcal infection according to the laboratory test results of symptoms, physical symptoms, gonococcus smear, culture, etc.
* Subjects having clinical suspicion of a gonococcal infection must have both of the following risk factors:once used three generations of cephalosporin invalid, and sensitive to this product (including gonorrhea urethritis, cervicitis, proctitis, pharyngitis).
* Male and female subject must agree to use contraception (male condoms) during intercourse from the Baseline Visit through completion of the TOC Visit.

Exclusion Criteria:

* Subject has a history of sensitivity to the study treatments, or components thereof, or a history of a drug (including erythromycin and any macrolide or ketolide drug) or other allergy that, in the opinion of the investigator or medical monitor, contraindicates his or her participation
* Subject has received any cephalosporinl therapy for the treatment of a gonococcal infection
* Pregnant or lactating women, or women Subject of childbearing age who were unwilling or unable to use acceptable methods of contraception throughout the study period.
* Famale subject who were positive for pregnancy tests at the time of inclusion or before the start of study drug use.
* Subject has risk of potentially serious drug interactions
* Subject has major diseases such as cardiovascular disease, hepatorenal disease and mental disease, or other factors, the researcher should not participate in the study according to comprehensive judgment
* Subject has a known history of alcohol or drug abuse
* Subject has a known any complicated or systemic gonorrhea infection, such as pelvic inflammatory disease, arthritis, endocarditis

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-07-03 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
bacterial eradicatio | Up to Day 8
  Number of subjects with culture-confirmed bacterial eradication of Neisseria gonorrhoeae from the urogenital site at the Test-of-Cure (TOC)

SECONDARY OUTCOMES:
clinical cure | Up to Day 8
  Number of subjects with disappearance of clinical symptoms and signs at the Test-of-Cure (TOC)
Comprehensive curative effect | Up to Day 8
  Number of subjects with culture-confirmed bacterial eradication of Neisseria gonorrhoeae from the urogenital site and disappearance of clinical symptoms and signs

CONTACTS AND LOCATIONS:
Overall Officials: pingyu P Zhou, Doctor, Principal Investigator — Shanghai Dermatology Hospital; shunming S Xu, Doctor, Principal Investigator — People's Hospital of Shanghai Pudong New Area; yanyue Tong, Doctor, Principal Investigator — People's Hospital of Quzhou; zhehu Jin, Doctor, Principal Investigator — The Affiliated Hospital of Yanbian University; bo Cheng, Doctor, Principal Investigator — First Affiliated Hospital of Fujian Medical University; wuqing W Wang, Doctor, Principal Investigator — The Central Hospital of Shanghai Minhang District; ping Wang, Doctor, Principal Investigator — The Third People's Hospital of Hangzhou

IPD SHARING:
Plan to Share IPD: No